CLINICAL TRIAL: NCT04922814
Title: Comparison for the Effect of Neuromuscular Blocking Agents Versus Sedation Alone on Severe ARDS Patients Due to COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman Abd El-Khalek Mohammed Glala, Principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Covid-19 ICU
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Sedation Complication; ICU Acquired Weakness
MeSH Terms: interventions — Muscle Relaxation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group(group A) (No Intervention): Only sedation for mechanically ventilated COVID patients
- Muscle relaxant group(group B) (Experimental): They will receive muscle relaxation treatment for at least 48 hours. Cisatracurium will be given. Short term infusions up to 24 hours will be given in a dose rate of 2-3 mic/Kg/min followed by intervallic shots of 2-5 mg.
  Interventions: Drug: muscle relaxation

INTERVENTIONS:
Drug: muscle relaxation — They will receive muscle relaxation treatment for at least 48 hours. Cisatracurium will be given. Short term infusions up to 24 hours will be given in a dose rate of 2-3 mic/Kg/min followed by intervallic shots of 2-5 mg.
  Arms: Muscle relaxant group(group B)

SUMMARY:
Many questions about management of COVID-19 are still not answered. So, we recruit this study aiming to evaluate improvement of oxygenation in COVID-19 patients with severe ARDS, to improve morbidity and mortality of ICU covid patients, to participate in understanding of real hidden pathophysiology of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Severe ARDS: PaO2/FiO2 <200, resistant hypoxemia and tachypnoea (RR > 40 breath/minute)
* Not relieved by high frequency nasal canula or CPAP.
* Need for invasive mechanical ventilation (uncooperative)

Exclusion Criteria:

* Patient relatives' refusal
* Not mechanically ventilated.
* Combination of female, corticosteroids administration and vecuronium muscle relaxant.
* Neuromuscular diseases (especially demyelinating diseases).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 | 48 hours
  ratio of arterial oxygen pressure in millilitre mercury to fraction of inspired oxygen at same time within the arterial blood gas

SECONDARY OUTCOMES:
Change in lung mechanics | 48 hours
  measurement of peak and plateau pressures in cm H2O, airway resistance in cm H2O. s/mL, static and dynamic compliance in Litre/cm H2O and positive end expiratory pressure in cm H2O from ventilator settings
SOFA score | 48 hours
  Fulfilment of modified SOFA (Sepsis Organ Failure Assessment) score sheet
Measurement of tissue perfusion | 48 hours
  Measurement of tissue perfusion by serum lactate in mmol/L and jugular venous oxygen saturation % from a sample withdrawn from CVP
Monitoring of Alveolar - Arterial Oxygen difference | 48 hours
  An arterial canula is to be introduced and a quantity of 0.5 ml of blood samples are obtained from radial artery and arterial blood gas analysis are performed after anti-coagulation by heparin. Alveolar-arterial oxygen tension difference:
  [P(A-a) DO2] = [(Pa-PH2O) × FiO2%-PaCO2-PaO2]
  * [(760-47) × FiO2%-PaCO2-PaO2]
  * [713 × FiO2%-PaCO2-PaO2]
28 days survival | after 28 days
  28 days survival
Recording risk factors | 28 days
  Recording risk factors as diabetes, renal failure, immunosuppression, smoking, COPD and obesity
Recording complications | 28 days
  Recording complications as VAP, HAP, neuromuscular weakness

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, faculty of medicine, anesthesia and ICU and pain management department, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Mason RJ. Pathogenesis of COVID-19 from a cell biology perspective. Eur Respir J. 2020 Apr 16;55(4):2000607. doi: 10.1183/13993003.00607-2020. Print 2020 Apr. PMID 32269085
- [Result] Neto AS, Pereira VG, Esposito DC, Damasceno MC, Schultz MJ. Neuromuscular blocking agents in patients with acute respiratory distress syndrome: a summary of the current evidence from three randomized controlled trials. Ann Intensive Care. 2012 Jul 26;2(1):33. doi: 10.1186/2110-5820-2-33. PMID 22835162
- [Result] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Derived] Hohmann F, Wedekind L, Grundeis F, Dickel S, Frank J, Golinski M, Griesel M, Grimm C, Herchenhahn C, Kramer A, Metzendorf MI, Moerer O, Olbrich N, Thieme V, Vieler A, Fichtner F, Burns J, Laudi S. Early spontaneous breathing for acute respiratory distress syndrome in individuals with COVID-19. Cochrane Database Syst Rev. 2022 Jun 29;6(6):CD015077. doi: 10.1002/14651858.CD015077. PMID 35767435